CLINICAL TRIAL: NCT04104269
Title: Comparative Risk Factors of Mechanical Structure Complications After Acute Myocardial Infarction
Brief Title: Mechanical Structure Complications After Acute Myocardial Infarction
Acronym: MSC-AMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Principal Investigator, Yan Wang, Ph D, FACC, Xiamen Cardiovascular Hospital, Xiamen University
Other Study IDs: 9215443687
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Heart rupture; Acute myocardial infarction
MeSH Terms: conditions — Heart Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mechanical Complications: Include free wall ventricular rupture and ventricular septal rupture
  Interventions: Diagnostic Test: Heart rupture
- Non-Mechanical Complications: Mechanical complications were not included in patients with AMI

INTERVENTIONS:
Diagnostic Test: Heart rupture — Free wall rupture and Ventricular septal rupture
  Groups: Mechanical Complications

SUMMARY:
To determine the incidence and factors associated with heart rupture (HR) in acute myocardial infarction patients.

DETAILED DESCRIPTION:
We compared characteristics and angiographic patterns of heart rupture and without heart rupture patients enrolled in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients be admitted for acute myocardial infarction (STEMI or NSTEMI)

Exclusion Criteria:

1. Non-cardiovascular comorbidity for AMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population of acute myocardial infarction (STEMI or NSTEMI) patients.
Sampling Method: Non-Probability Sample
Enrollment: 35621 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Heart rupture | Mortality 30 days
  Includee free wall ventricular rupture and ventricular septal rupture

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, PhD, Study Chair — Xiamen Cardiovascular Hospital, Xiamen University
Locations (1):
- Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No